CLINICAL TRIAL: NCT05050422
Title: The Effects of Trunk Impairment on Fatigue and Balance in Children With CP
Brief Title: The Effects of Trunk Impairment on Fatigue and Balance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Mehmet Duray, Principal Investigator, Suleyman Demirel University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: E-60116787-020-67242
Record Dates: First submitted 2021-09-13; First posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator)
  Interventions: Diagnostic Test: Trunk Impairment Scale (TIS), PedsQLTM Multidimensional Fatigue Scale (PedsQL-MFS), Pediatric Balance Scale (PBS)
- Study (Active Comparator)
  Interventions: Diagnostic Test: Trunk Impairment Scale (TIS), PedsQLTM Multidimensional Fatigue Scale (PedsQL-MFS), Pediatric Balance Scale (PBS)

INTERVENTIONS:
Diagnostic Test: Trunk Impairment Scale (TIS), PedsQLTM Multidimensional Fatigue Scale (PedsQL-MFS), Pediatric Balance Scale (PBS) — control/study group

SUMMARY:
Fatigue is a common symptom associated with cerebral palsy (CP); it has been estimated that up to 40% of adolescents with CP experience fatigue that impacts their quality of life and daily activities. Although fatigue was stated as the primary symptom, a limited number of studies were found on secondary motor and nonmotor symptoms related to trunk control in children when the literature was examined.

ELIGIBILITY:
Inclusion Criteria:

aged between 2-18 years old; (2) had a form of CP; (3) had the cognitive competence to participate to the all assessments.

Exclusion Criteria:

The sufferers who had an additional neurological or musculoskeletal disability, unstable medical conditions, any recent medical intervention (such as tendon lengthening surgery or botulinum toxin injection…) were excluded

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-09-13 (Estimated); Primary Completion 2021-10-13 (Estimated); Study Completion 2021-10-13 (Estimated)

PRIMARY OUTCOMES:
Trunk Impairment Scale (TIS) | 1 month
PedsQLTM Multidimensional Fatigue Scale (PedsQL-MFS) | 1 month
Pediatric Balance Scale (PBS) | 1 month

IPD SHARING:
Plan to Share IPD: Undecided